CLINICAL TRIAL: NCT04559971
Title: A Randomised, Double-blind, Placebo-controlled Phase 1 Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneously Administered SLN124 in Healthy Volunteers
Brief Title: A Phase 1 Study to Evaluate the Safety, Tolerability, PK and PD of SLN124 in Healthy Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Silence Therapeutics plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SLN124-003
Record Dates: First submitted 2020-09-08; First posted 2020-09-23 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1.0mg/kg (Experimental): Drug: SLN124
  Interventions: Drug: SLN124
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- 3.0mg/kg (Experimental): Drug: SLN124
  Interventions: Drug: SLN124
- Optional Cohort (Experimental): An additional dose level may be explored
  Interventions: Drug: SLN124

INTERVENTIONS:
Drug: SLN124 — SLN124 for subcutaneous (s.c.) injection
  Arms: 1.0mg/kg; 3.0mg/kg; Optional Cohort
Drug: Placebo — Sodium chloride for s.c. injection
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and tolerability of SLN124 in healthy volunteers.

DETAILED DESCRIPTION:
This first-in-human (FIH) study will investigate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of SLN124 after single ascending s.c. doses in healthy male and female subjects.

Up to 3 cohorts of 24 healthy volunteers will be enrolled. Each subject will receive a single dose of SLN124 or placebo given by subcutaneous (s.c) injection.

ELIGIBILITY:
Inclusion Criteria:

* Normotensive male or female volunteers, with a body mass index of 18.0-30.0 kg/m2.
* Deemed healthy on the basis of a clinical history, physical examination, ECG, vital signs, and laboratory tests of blood and urine.
* Agree to follow the contraception requirements of the trial.
* Able to give fully informed written consent.
* Agree not to donate blood or blood products during the study and for up to 3 months after the administration of the trial medication.

Exclusion Criteria:

* History or presence of iron deficiency or iron deficiency anaemia and/or currently receiving oral or parenteral iron supplementation as treatment for those conditions.
* Positive tests for hepatitis B & C, HIV
* Drug or alcohol abuse.
* Smoke more than 10 cigarettes (or equivalent) daily.
* Use of over-the-counter medication (with the exception of paracetamol [acetaminophen]) during the 7 days before the first dose of trial medication, or prescribed medication (with the exception of hormone replacement therapy [HRT]) during the 28 days before first dose of trial medication.
* Use of supplement(s) during the 28 days before screening.
* Participation in other clinical trials of unlicensed medicines, or loss of more than 400 mL blood, within the previous 3 months.
* Clinically relevant abnormal medical history or concurrent medical condition.
* Pre-menopausal females who are pregnant or lactating, or who are sexually active and not using a reliable method of contraception.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | 8 weeks
  safety and tolerability

SECONDARY OUTCOMES:
Pharmacokinetic: peak plasma concentration (Cmax) | 7 days
Pharmacokinetic: area under the plasma concentration (AUC) | 7 days
Pharmacokinetic: apparent total clearance from plasma after s.c injection (CL/F) | 7 days

OTHER OUTCOMES:
Pharmacodynamic: change in ferritin | 8 weeks
Pharmacodynamic: change in TSAT | 8 weeks
Pharmacodynamic: change in hepcidin | 8 weeks
Pharmacodynamic: change in haemoglobin | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Giles Campion, MD, Study Director — Silence Therapeutics
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom

REFERENCES:
- [Derived] Porter JB, Scrimgeour A, Martinez A, James L, Aleku M, Wilson R, Muckenthaler M, Boyce M, Wilkes D, Schaeper U, Campion GV. SLN124, a GalNAc conjugated 19-mer siRNA targeting tmprss6, reduces plasma iron and increases hepcidin levels of healthy volunteers. Am J Hematol. 2023 Sep;98(9):1425-1435. doi: 10.1002/ajh.27015. Epub 2023 Jul 27. PMID 37497888